CLINICAL TRIAL: NCT00873132
Title: BTC Neuropsychological Database:Prospective Study
Brief Title: BTC Neuropsychological Database
Status: Withdrawn | Type: Observational
Why Stopped: No Funding
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00012450
Record Dates: First submitted 2009-03-30; First posted 2009-04-01 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Data Collection: Collect data both retrospectively and prospectively on subjects seen at the Preston Robert Tisch Brain Tumor Center

SUMMARY:
Purpose and Objective:

The purpose of this study is to collect data both retrospectively and prospectively, by consent, on subjects seen in the PRTBTC. This information will be useful to the investigators to generate hypotheses for planning further psychosocial and medication intervention studies that will hopefully improve primary brain tumor patients' QOL.

DETAILED DESCRIPTION:
Study Activities and Population Group:

Retrospective dates will be 3/1/06 through the approval date for the prospective component of this study. The data will be neurocognitive, depression, tumor-related, overall quality of life (QOL), treatment, and demographic variables. The investigators research aims are to

* compute correlations among these different variables
* to test significant predictors of QOL. The investigators also will conduct a retrospective review of all brain tumor patients evaluated at the neuropsychology clinic at the PRT-BTC from the date that this prospective study is approved back to 3/20/2006.

Data Analysis and Risk/Safety Issues:

The medical record review does not present any obvious source of risk or discomfort to patients and their families. For both the retrospective and prospective components of the study, as the data for the proposed study were already collected as a part of the standard of care at the Preston Robert Tisch Brain Tumor Center at Duke, there are no additional risks to the study sample as a result of data collection.

ELIGIBILITY:
Inclusion Criteria:

* Data collected both retrospectively and prospectively, by consent, on subjects with brain tumors seen in the Preston Robert Tisch Brain Tumor Center (PRTBTC).
* Retrospective dates will be 3/1/06 through the approval date for the prospective component of this study.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For those patients enrolled, we will conduct analysis on data that is gathered during neuropsychological testing visits to better describe the pattern of neurocognitive deficits typically seen in our patient population and to publish our findings with the goal of informing a larger scientific community.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Bivariate correlational analyses will be conducted to examine associations between neuropsychological, depression, demographic, medication data tumor-related treatment , and QoL variables. | 5years

SECONDARY OUTCOMES:
In exploratory analyses, FACT-BR scale scores will be regressed on candidate neurocognitive predictors while controlling for other potentially confounding variables using hierarchical regression analyses. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Renee Raynor, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States